CLINICAL TRIAL: NCT05254249
Title: Analysis of Gut Microbiota, Psoriasis Area and Severity Index, Interleukin-17, Tumor Necrosis Factor -α, Interleukin-10, and Foxp3 in Psoriasis Vulgaris After Supplementation With Lactobacillus Plantarum IS-10506
Brief Title: Clinical Trial of Probiotic Supplementation in Psoriasis Vulgaris
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Soetomo General Hospital (Other Government)
Collaborators: Universitas Airlangga (Other)
Responsible Party: Principal Investigator, Menul Ayu Umborowati, dr., Sp.KK, doctor, dermatovenereologist, Dr. Soetomo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0315/KEPK/XI/2021
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Psoriasis Vulgaris
Keywords: Psoriasis Vulgaris; Psoriasis Area and Severity Index; Interleukin-17; Tumor Necrosis Factor- A; Interleukin-10; Foxp3; Lactobacillus Plantarum IS-10506; Gut Microbiota
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: A double blinded randomized clinical trial using a prospective cohort method in psoriasis vulgaris patients with purposive sampling.
Who Masked: Participant, Investigator
Masking Description: Probiotic and placebo packaging are made the same, and drug code is randomized by pharmacy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group (Active Comparator): In the treatment group, intervention was given in the form of standard therapy and probiotic Lactobacillus plantarum IS 10605 in the amount of 2x1010 CFU for 12 weeks.
  Interventions: Drug: Lactobacillus Plantarum IS-10506
- Placebo Group (Placebo Comparator): In the placebo group, intervention was given in the form of standard therapy and placebo 2x1 sachets for 12 weeks.
  Interventions: Other: Placebo
- Healty Control Group (No Intervention): Healthy control group was not given any treatment. Stool samples were taken to examine the gut microbiota profile.

INTERVENTIONS:
Drug: Lactobacillus Plantarum IS-10506 — Indonesian original probiotic, given in capsule form with a dose of 2 x 1010 CFU
  Other Names: Probiotic
  Arms: Treatment Group
Other: Placebo — Placebo is an empty drug, given in capsule form with a dose of 2x1 sachets
  Arms: Placebo Group

SUMMARY:
Psoriasis is a chronic inflammatory skin disease (chronic and recurrent) which is influenced by various factors, namely genetics, immunological processes, and environmental triggers such as infection, obesity, smoking, and drugs.

The provision of probiotic Lactobacillus plantarum IS-10506, an Indonesian original probiotic strain, is expected to be an effective, safe, and affordable alternative for psoriasis treatment for psoriasis patients in Indonesia.

This study aimed to evaluate changes in gut microbiota profile, cytokines IL-17, TNF-a, IL-10, Foxp3, and disease severity of psoriasis vulgaris patients after supplementation with Lactobacillus plantarum IS-10506. The results of this study are expected to be the basis for the use of Lactobacillus plantarum IS-10506 in the therapy of psoriasis vulgaris which is included in the Clinical Practice Guide in Indonesia, which will ultimately help improve the quality of life of psoriasis patients.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory skin disease (chronic and recurrent) which is influenced by various factors, namely genetics, immunological processes, and environmental triggers such as infection, obesity, smoking, and drugs. Psoriasis can increase the incidence of other diseases such as joint disorders, cardiovascular disorders, and psychological. Symptoms of psoriasis on the skin are red, well-defined plaques covered with thick, white, layered scales. The incidence of psoriasis is quite large, known to affect 0.09 - 11.4% of the world's population with rates varying between regions. Data in Indonesia is estimated that there are 2-6 million psoriasis sufferers in 2010, with a prevalence range of 1-3% in several teaching hospitals. During the period from 2016 to 2018, psoriasis vulgaris patients in the outpatient unit of RSUD Dr. Soetomo Surabaya recorded as many as 208 or 0.46% of all skin patients.

One of the mechanisms of psoriasis is abnormalities in Treg cells (cells that play a role in expressing Foxp3), resulting in an imbalance in the immune system with the dominance of T helper 1 (Th1) and T helper 17 (Th17) cells. In addition, the composition of the gut microbiota (collection of bacteria) in psoriasis patients is different from that of healthy people. The composition of the gut microbiota can be influenced by race, geography, and eating habits. Until now there has been no report on the intestinal microbiota profile of psoriasis patients in Indonesia.

The provision of probiotic Lactobacillus plantarum IS-10506, is expected to be an effective, safe, and affordable alternative for psoriasis treatment for psoriasis patients in Indonesia. Lactobacillus plantarum IS-10506 is produced from Dadih, a traditional fermented milk from West Sumatra, Indonesia. This probiotic is expected to be most compatible with the composition of the gut microbiota of Indonesians because it comes from an environment with similar exposure to pathogenic bacteria.

This study aimed to evaluate changes in gut microbiota profile, cytokines IL-17, TNF-a, IL-10, Foxp3, and disease severity of psoriasis vulgaris patients after supplementation with Lactobacillus plantarum IS-10506. The results of this study are expected to be the basis for the use of Lactobacillus plantarum IS-10506 in the therapy of psoriasis vulgaris which is included in the Clinical Practice Guide in Indonesia, which will ultimately help improve the quality of life of psoriasis patients.

ELIGIBILITY:
Inclusion Criteria:

Patient Group Inclusion Criteria:

1. Psoriasis vulgaris patients with or without treatment
2. Mild to moderate degree
3. Age 18-70 years old
4. Willing to give informed consent

Healthy Control Group Inclusion Criteria:

1. Undiagnosed as Psoriasis
2. Body mass index (BMI) is matched with the patient group
3. Age 18-70 years old
4. Willing to give Informed Consent

Exclusion Criteria:

Patient Group Exclusion Criteria:

1. Patients on systemic treatment with corticosteroids, methotrexate, cyclosporine, or biologic agents within 3 months prior to sampling
2. Take oral antibiotics, laxatives, and proton pump inhibitors (PPI) within 14 days before stool sampling
3. Suffering from severe systemic disease, diarrhea
4. Pustular psoriasis patients
5. Take probiotics within 30 days before stool sampling

Healthy Control Group Exclusion Criteria:

1. Patients on systemic treatment with corticosteroids, methotrexate, cyclosporine, or biologic agents within 3 months before stool sampling
2. Take oral antibiotics, laxatives, and proton pump inhibitors (PPI) within 14 days before stool sampling
3. Suffering from severe systemic disease, diarrhea

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Alpha and beta | 12 weeks
  Alpha and beta diversity in gut microbiota profiles
Serum levels | 12 weeks
  Changes in serum levels of TNF-α, IL-17, IL-10, and Foxp3 by ELISA method
PASI scores | 12 weeks
  Changes in PASI scores after the intervention

SECONDARY OUTCOMES:
DLQI | 12 weeks
  Changes in the score of impaired quality of life due to skin diseases experienced using the DLQI questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Menul Ayu Umborowati, Specialist, Study Chair — Dr. Soetomo General Hospital
Locations (1):
- Universitas Airlangga, Surabaya, East Java, Indonesia